CLINICAL TRIAL: NCT02283333
Title: Treatment of Prolonged Grief Disorder in Combat Veterans
Acronym: PGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLNA-001-14S; CX001102 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2014-10-23; First posted 2014-11-05 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Prolonged Grief Disorder
Keywords: Behavioral Activation; Therapeutic Exposure; Mental Health; Veterans; Complicated Grief; Military; Treatment; Cognitive Therapy; Bereavement; Complicated Bereavement
MeSH Terms: conditions — Prolonged Grief Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BATE-G (Experimental): Behavioral Activation and Therapeutic Exposure - Grief therapy are delivered in 7 weekly sessions to the participant.
  Interventions: Behavioral: BATE-G
- Standard Treatment (Active Comparator): Cognitive Restructuring and Supportive Grief Counseling are delivered in 7 weekly sessions to the participant.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: BATE-G — Behavioral Activation and Therapeutic Exposure - Grief therapy is delivered in 7 weekly sessions to the participant.
  Arms: BATE-G
Behavioral: Standard Treatment — Cognitive Restructuring and Supportive Grief Counseling is delivered in 7 weekly sessions to the participant.
  Arms: Standard Treatment

SUMMARY:
The purpose of this study is to compare the efficacy of an experimental treatment (termed BATE-G) for Prolonged Grief Disorder (PGD) in Veterans compared to the current, VA-approved standard of care treatment. Currently, treatments for grief in Veterans remain understudied. Our research group has recently completed pilot work on an innovative, technology-leveraged treatment protocol for PGD that combines Behavioral Activation with Therapeutic Exposure (BATE) and appears readily applicable to the Veteran and Military populations. Per the VA / DoD Iraq War Clinician Guide, 2nd ed., the current standard of treatment is Cognitive Restructuring and Supportive Grief Counseling.

The study will enroll 140 Veterans, aged 21 years and older, who served in any combat era. All Veterans will meet criteria for PGD. There will be assessments at baseline, 1 week, 3 months, and 6 months post treatment. During the treatment phase, Veterans will undergo 7 weekly sessions of either BATE-G or standard treatment. Sessions 2-6 will be delivered via televideo to the Veteran's home.

We hypothesize that BATE-G will be more effective than standard treatment in reducing symptoms of PGD, both at post-treatment and follow-up. Moreover, BATE-G will be more effective in reducing acute emotional distress and preventing long-term emotional distress in terms of general depression and anxiety symptoms. BATE-G will result in increased frequency of completed positively reinforcing, community-based events when compared to Cognitive Restructuring and Supportive Grief Counseling. BATE-G will also result in greater improvements in perceived social support and health.

Note: This project is the first evidence-based treatment for PGD in military populations, thus addressing a significant service gap.

DETAILED DESCRIPTION:
The 'dual burden' of (a) loss of a fellow service member in the context of (b) experiencing repeated extreme life threat is unique to military combat personnel and a core characteristic of combat-related Prolonged Grief Disorder (PGD), a disorder as prevalent as Post-traumatic stress disorder and associated with functional impairment, disability, and suicidality. Effective treatments for depression and PTSD have proven less than adequate in treating PGD when each is offered in isolation; and simply combining these 12-16 week treatment regimens into a 24-36 week treatments is not a viable approach, particularly with a population predisposed to avoiding extended mental health care. This project addresses the need for a Veteran/ military specific treatment of PGD, and uses technology to deliver this treatment in a format that is far more likely to be accepted by military personnel and Veterans. This study will impact clinical practice by providing the first evidence for effective treatment of PGD in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be either Active Duty Service Personnel/Veterans of any service era.
* Participants may be male or female,

  * age 21 and above,
  * with a diagnosis of Prolonged Grief Disorder.
* Veterans starting a new psychotropic medication at baseline will be asked to wait 4 weeks for medication stabilization before starting the study.

Exclusion Criteria:

* Actively psychotic or demented persons,
* Individuals with both suicidal ideation and clear intent,
* Individuals with homicidal ideation and or intent,
* Individuals meeting criteria for substance dependence,
* Individuals who cannot or are unwilling to schedule regular weekly appointments (with the exception of Veterans who have medical and/or transportation barriers,
* Individuals who are already enrolled in another trial for PTSD and/or depression will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron E. Acierno, PhD MS BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BATE-G | Standard Treatment
Started | 77 | 78
Completed | 63 | 64
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BATE-G | Standard Treatment | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 65 | 135
  >=65 years | 7 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.01 (12.24) | 47.35 (13.13) | 46.68 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 61 | 65 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 70 | 74 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 42 | 45 | 87
  White | 24 | 28 | 52
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77 | 78 | 155

OUTCOME MEASURES:

1. Primary Outcome: Inventory of Complicated Grief - Revised (ICG-R)
Description: The Inventory of Complicated Grief (ICG) Revised is a self-report instrument that allows for the dimensional assessment of the severity of complicated grief symptoms. It has 34 items with scores ranging from 30 to 150. Min score 50; max score 143 indicated at baseline. Higher scores indicate worse outcomes.
Time Frame: Baseline
Population: Veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 93.15 (19.79) | 93.10 (21.59)

2. Primary Outcome: Inventory of Complicated Grief - Revised (ICG-R)
Description: The Inventory of Complicated Grief (ICG) is a self-report instrument that allows for the dimensional assessment of the severity of complicated grief symptoms. It has 34 items with scores ranging from 30 to 150. Min score 33.31; max score 133 indicated at post. Higher scores indicate worse outcomes.
Time Frame: 8 weeks
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 78.8 (19.4) | 78.6 (21.2)

3. Primary Outcome: Inventory of Complicated Grief - Revised (ICG-R)
Description: The Inventory of Complicated Grief (ICG) is a self-report instrument that allows for the dimensional assessment of the severity of complicated grief symptoms. It has 34 items with scores ranging from 30 to 150. Min score 31.97; max score 150 indicated at 3 month. Higher scores indicate worse outcomes.
Time Frame: 3 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 79.4 (22.7) | 81.4 (22.8)

4. Primary Outcome: Inventory of Complicated Grief - Revised (ICG-R)
Description: The Inventory of Complicated Grief (ICG) is a self-report instrument that allows for the dimensional assessment of the severity of complicated grief symptoms. It has 34 items with scores ranging from 30 to 150. Min score 30; max score 141 indicated at 6 month. Higher scores indicate worse outcomes.
Time Frame: 6 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 78.6 (22.9) | 80.0 (21.4)

5. Secondary Outcome: Beck Depression Inventory - II (BDI-II)
Description: Beck Depression Inventory-II is a 21 item measure of depressive severity with scores ranging from 0 to 63. Min score 0; max score 61 indicated at baseline. Higher scores indicate worse outcomes.
Time Frame: Baseline
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 28.5 (11.8) | 28.8 (14.0)

6. Secondary Outcome: PTSD Checklist for DSM-5 (PCL 5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD with scores ranging from 0 to 80. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Min score 2; max score 76 indicated at baseline. Higher scores indicate worse outcomes.
Time Frame: Baseline
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 48.0 (15.1) | 46.2 (16.5)

7. Secondary Outcome: Beck Depression Inventory - II (BDI-II)
Description: Beck Depression Inventory-II is a 21 item measure of depressive severity with scores ranging from 0 to 63. Min score 0; max score 58 indicated at post. Higher scores indicate worse outcomes.
Time Frame: 8 weeks
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 23.0 (11.6) | 22.1 (10.9)

8. Secondary Outcome: Beck Depression Inventory - II (BDI-II)
Description: Beck Depression Inventory-II is a 21 item measure of depressive severity with scores ranging from 0 to 63. Min score 0; max score 52 indicated at 3 month. Higher scores indicate worse outcomes.
Time Frame: 3 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 22.0 (10.5) | 22.2 (11.2)

9. Secondary Outcome: Beck Depression Inventory - II (BDI-II)
Description: Beck Depression Inventory-II is a 21 item measure of depressive severity with scores ranging from 0 to 63. Min score 0; max score 58 indicated at 6 month. Higher scores indicate worse outcomes.
Time Frame: 6 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 21.1 (11.2) | 23.4 (11.3)

10. Secondary Outcome: PTSD Checklist for DSM-5 (PCL 5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD with scores ranging from 0 to 80. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Min score 0; max score 72 indicated at post. Higher scores indicate worse outcomes.
Time Frame: 8 weeks
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 34.5 (15.8) | 33.9 (16.5)

11. Secondary Outcome: PTSD Checklist for DSM-5 (PCL 5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD with scores ranging from 0 to 80. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Min score 0; max score 76 indicated at 3 month. Higher scores indicate worse outcomes.
Time Frame: 3 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 35.3 (16.8) | 37.6 (16.3)

12. Secondary Outcome: PTSD Checklist for DSM-5 (PCL 5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD with scores ranging from 0 to 80. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Min score 0; max score 76 indicated at 6 month. Higher scores indicate worse outcomes.
Time Frame: 6 months
Population: veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BATE-G | Standard Treatment
Number analyzed (Participants) | 77 | 78
score on a scale | 33.3 (16.7) | 36.0 (14.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 5 years, 1 month.
Description: Adverse events and serious adverse events were recorded in accordance with clinicaltrials.gov definitions.
Arm/Group | BATE-G | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/78
Other Adverse Events (participants affected / at risk) | 0/77 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BATE-G (N=77) | Standard Treatment (N=78)
Serious Adverse Event (Psychiatric disorders) | 0 | 1 — Participant attempted suicide by attempting to overdose on blood pressure medication pills.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02283333/Prot_SAP_000.pdf